CLINICAL TRIAL: NCT00563069
Title: Premedication With Oral Midazolam in Patients Undergoing Rigid Cystoscopy: A Randomized, Double-blind, Placebo-controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CRE-2005.250-T; HARECCTR0500009
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Cystoscopy
Keywords: diagnostic and therapeutic rigid cystoscopy
MeSH Terms: conditions — Disease | interventions — Midazolam

INTERVENTIONS:
Drug: Midazolam

SUMMARY:
To investigate the efficacy of oral midazolam for patients undergoing rigid cystoscopy in:

1. relieving patient's anxiety and improving satisfaction
2. reducing procedure-related pain
3. facilitating the diagnostic and therapeutic interventions during rigid cystoscopy

ELIGIBILITY:
Inclusion Criteria:

* Elective rigid cystoscopy
* Either diagnostic or therapeutic
* Age between 18 to 80

Exclusion Criteria:

* Patients with allergy to midazolam or other benzodiazepine groups
* Pregnancy
* Emergency rigid cystoscopy
* ASA class 3 or above
* Patients on psychiatric medications
* Alcoholics

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-09; Study Completion 2006-12 (Estimated)

PRIMARY OUTCOMES:
Pain score during the procedure as assessed by visual analog scale

SECONDARY OUTCOMES:
Patient's satisfaction
Patient's willingness to repeat the procedure
Patient's cooperativeness during the procedure as assessed by surgeons

CONTACTS AND LOCATIONS:
Overall Officials: Shirley YW Liu, Dr, Principal Investigator — Department of Surgery, Prince of Wales Hospital/ The Chinese Univerisity of Hong Kong
Locations (1):
- Department of Surgery, Prince of Wales Hospital, Hong Kong, China